CLINICAL TRIAL: NCT02075476
Title: Prospective, Randomized and Double Blind Study of Parallels Groups for Evaluating the Effectiveness Between Two Surgical Techniques for Reconstruction of Humeral Proximal Extremity Fractures in Three or Four Fragments
Brief Title: Effectiveness Between Two Surgical Techniques for Reconstruction of Humeral Proximal Extremity Fractures
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Carlos Alvarez (Other)
Responsible Party: Sponsor-Investigator, Carlos Alvarez, Head of Department, Hospital General Universitario Gregorio Marañon
Organization: Hospital General Universitario Gregorio Marañon (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: FRALUX-34
Record Dates: First submitted 2014-02-06; First posted 2014-03-03 (Estimated); Results first posted 2020-04-14 (Actual); Last update posted 2020-04-14 (Actual); Status verified 2020-04

CONDITIONS: A02.835.232.087.090.400.400
Keywords: Fracture-luxation; humeral proximal extremity; Hemiarthroplasty; reverse Arthroplasty
MeSH Terms: interventions — Hemiarthroplasty

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Hemiarthroplasty Global Fx(DePuy) (Active Comparator): in this technique the prosthesis is implanted in similar approach to shoulder anatomy
  Interventions: Procedure: Hemiarthroplasty
- reverse arthroplasty Delta Xtent(DePuy) (Experimental): In this technique the prosthesis is implanted in the inverse mode of shoulder anatomy
  Interventions: Procedure: reverse arthroplasty

INTERVENTIONS:
Procedure: Hemiarthroplasty
  Arms: Hemiarthroplasty Global Fx(DePuy)
Procedure: reverse arthroplasty
  Arms: reverse arthroplasty Delta Xtent(DePuy)

SUMMARY:
The purpose of this study is to evaluate the effectiveness and safety of two surgical techniques for the treatments of proximal extremity humeral fractures and fractures luxation in three o four fragments of Neer's classification.

DETAILED DESCRIPTION:
Proximal extremity humeral fractures present high prevalence. It's estimated about 10% of all fractures. Their incidence is 6,6/1000 people-year and this amount increases from 40 years old. The majority are successfully treated with immobilization and rehabilitation. The surgical treatment is recommended in case of displacement. In elderly population with fractures types three or four of Neer's classification there is no consensus on which technique is the best surgical option. Classically hemiarthroplasty has been widely performed as a reconstruction method but its outcomes in old patients are unclear due to the bad bone quality and joint features. Recently some authors recommend the reverse arthroplasty in patients over 70 years old . The aim of this study is to compare the results between Hemiarthroplasty and reverse arthroplasty in patients over 70 years old. As far as the investigators are concerned there's no published studies like this.

ELIGIBILITY:
Inclusion Criteria:

* Patients with humeral proximal extremity fracture or fracture luxation in three or four fragments of Neer's classification.
* Patient 70 years older
* Signed informed consent.

Exclusion Criteria:

* Any condition to make worse the functional recovery or avoid the patient collaboration with the rehabilitation program ( cognitive disability, neurological pathology…)

  * Glenohumeral osteoarthritis
  * Inflammatory arthropathies
  * Previous cuff arthropatyy
  * High surgical or anesthesia risk
  * Any disease or condition that the investigator finds decisive for exclusion.

Min Age: 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 40 (Actual)
Dates: Start 2013-05 (Actual); Primary Completion 2015-08-05 (Actual); Study Completion 2016-08-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Carlos Alvarez, MD, Principal Investigator — Hospital General Universitario Gregorio Marañon
Locations (1):
- Hospital General Universitario Gregorio Marañon, Madrid, Spain

REFERENCES:
- [Derived] Handoll HH, Elliott J, Thillemann TM, Aluko P, Brorson S. Interventions for treating proximal humeral fractures in adults. Cochrane Database Syst Rev. 2022 Jun 21;6(6):CD000434. doi: 10.1002/14651858.CD000434.pub5. PMID 35727196

RESULTS

PARTICIPANT FLOW:
Groups:
- Hemiarthroplasty Global Fx(DePuy): in this technique the prosthesis is implanted in similar approach to shoulder anatomy
  Hemiarthroplasty
- Reverse Arthroplasty Delta Xtent(DePuy): In this technique the prosthesis is implanted in the inverse mode of shoulder anatomy
  reverse arthroplasty
Period: Overall Study
Arm/Group | Hemiarthroplasty Global Fx(DePuy) | Reverse Arthroplasty Delta Xtent(DePuy)
Started | 20 | 20
Completed | 17 | 15
Not Completed | 3 | 5
Not completed — Death | 2 | 2
Not completed — Lost to Follow-up | 1 | 3

BASELINE CHARACTERISTICS:
Population: All patients 70 years of age or older with 3- or 4-part shoulder fractures were included in the study
Groups:
- Total: Total of all reporting groups
Arm/Group | Hemiarthroplasty Global Fx(DePuy) | Reverse Arthroplasty Delta Xtent(DePuy) | Total
Number analyzed (Participants) | 20 | 19 | 39
Age, Continuous [Mean (Full Range); unit: years] | 76 [71 to 85] | 77 [71 to 85] | 76 [71 to 85]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14 | 13 | 27
  Male | 6 | 6 | 12
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  Spain | 20 | 19 | 39

OUTCOME MEASURES:

1. Primary Outcome: Effectiveness Will be Measured for AMERICAN SHOULDER AND ELBOW (ASES) Score
Description: changes en ASES (AMERICAN SHOULDER AND ELBOW) score will be measured.
  The ASES questionnaire is composed of both a physician-rated component and a patient-reported component. The patient questions focus on joint pain, instability, and activities of daily living. This questionary includes a section on pain (7 items) and a section on activities of daily living (10 items). Scores range from 0 to 100 with a score of 0 indicating a worse shoulder condition and 100 indicating a better shoulder condition.
Time Frame: 36 months
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Hemiarthroplasty Global Fx(DePuy) | Reverse Arthroplasty Delta Xtent(DePuy)
Number analyzed (Participants) | 19 | 20
score on a scale | 66 [60 to 81] | 77 [72 to 85]
Statistical Analysis 1: Comparison: Hemiarthroplasty Global Fx(DePuy) vs Reverse Arthroplasty Delta Xtent(DePuy); Test type: Equivalence — Normality in sample distribution was tested using the Kolmororov-Smirnov test and graphic models. For descriptive variables we use Pearson's Chi-square, and for the study of numerical variables over time we use a mixed linear test; p = 0.048, Mixed Models Analysis

2. Primary Outcome: Effectiveness Will be Measured for Constant Score
Description: changes in Constant score will be measured.
  The Constant-Murley score (CMS) is a 100-points scale composed of a number of individual parameters. These parameters define the level of pain and the ability to carry out the normal daily activities of the patient. The Constant-Murley score was introduced to determine the functionality after the treatment of a shoulder injury.
  The test is divided into four subscales: pain (15 points), activities of daily living (20 points), strength (25 points) and range of motion: forward elevation, external rotation, abduction and internal rotation of the shoulder (40 points). The higher the score, the higher the quality of the function.
Time Frame: 36 months
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Hemiarthroplasty Global Fx(DePuy) | Reverse Arthroplasty Delta Xtent(DePuy)
Number analyzed (Participants) | 19 | 20
score on a scale | 53 [45 to 59] | 70 [65 to 80]
Statistical Analysis 1: Comparison: Hemiarthroplasty Global Fx(DePuy) vs Reverse Arthroplasty Delta Xtent(DePuy); Test type: Equivalence — [test comment as in outcome 1, analysis 1]; p = 0.001, Mixed Models Analysis

3. Primary Outcome: Effectiveness Will be Measured for DASH (Disabilities of the Arm, Shoulder and Hand) Score
Description: changes in DASH (Disabilities of the Arm, Shoulder and Hand) score will be measured.
  The Disabilities of the Arm, Shoulder and Hand (DASH) outcome measure is a 30-item, self-report questionnaire designed to assess the patient's health status during the previous week. The items enquire about the degree of difficulty in performing different physical activities because of arm, shoulder and hand problems (21 items), the severity of each of the symptoms of pain, activity-related pain, tingling, weakness and stiffness (five items) and the impact of the problem on social functioning, work, sleep and self-image (four items). Each item has five response options. The scores are then used to calculate a scale score ranging from 0 (no disability) to 100 (most severe disability)
Time Frame: 36 months
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Hemiarthroplasty Global Fx(DePuy) | Reverse Arthroplasty Delta Xtent(DePuy)
Number analyzed (Participants) | 19 | 20
score on a scale | 26 [13 to 33] | 13 [10 to 26]
Statistical Analysis 1: Comparison: Hemiarthroplasty Global Fx(DePuy) vs Reverse Arthroplasty Delta Xtent(DePuy); Test type: Equivalence — [test comment as in outcome 1, analysis 1]; p = 0.011, Mixed Models Analysis

ADVERSE EVENTS:
Time Frame: 36 months
Description: Patient follow-up was done in consultations through five successive visits, at 6 weeks, at 3 months, at 6 months, a year, and the final review (minimum 40 months). These reviews were carried out by a specialist who was unaware of the prosthetic model that patients were wearing. (Masking technique).
  As an adverse event we have collected the appearance of infections, instability or prosthetic loosening.
  No infections, instability or prosthetic loosening were reported in any patient.
Arm/Group | Hemiarthroplasty Global Fx(DePuy) | Reverse Arthroplasty Delta Xtent(DePuy)
All-Cause Mortality (participants affected / at risk) | 0/19 | 0/20
Serious Adverse Events (participants affected / at risk) | 0/19 | 0/20
Other Adverse Events (participants affected / at risk) | 0/19 | 0/20

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No